CLINICAL TRIAL: NCT04719338
Title: Occult Hepatitis C Virus Infection In Hemodialysis Patients Who Achieved A Sustained Virological Response To Directly Acting Antiviral Drugs: Is It A Concern ?
Brief Title: Occult HCV Infection After DAAD Treatment in Haemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, lecturer, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: occult HCV in dialysis
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Hepatitis C
Keywords: occult HCV, direct antiviral drugs, haemodialysis
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: This research is a cross sectional study. Target population: thirty patients with end-stage renal disease (ESRD) receiving hemodialysis treatment from different dialysis centers in Alexandria will be enrolled in the study after achieving sustained virological response 24 weeks after the end of treatment with directly acting antiviral drugs (DAADs).will be screened for the presence of occult HCV infection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): Immediately after confirmation of 24 weeks SVR after the end of treatment, we will collect samples of peripheral blood from each patient into EDTA tube and test for HCV RNA in peripheral blood mononuclear cells (PBMCs) .
  All patients included in this study will be subjected to full history taking and thorough clinical examination. The initial pre treatment data of the patients will be revised including body mass index (BMI), pre treatment status (naïve,experienced), pretreatment viral load by sensitive real-time HCV PCR technique, liver function tests, complete blood count, prothrombin time, international normalized ratio , Child-Pugh score, MELD score and FIB-4 score .
  Interventions: Diagnostic Test: presence of HCV RNA in peripheral blood mononuclear cells (PBMCs) .

INTERVENTIONS:
Diagnostic Test: presence of HCV RNA in peripheral blood mononuclear cells (PBMCs) . — samples of peripheral blood from each patient into EDTA tube will be collected and tested for HCV RNA in peripheral blood mononuclear cells (PBMCs) .
  Other Names: occult HCV infection

SUMMARY:
This research aims to evaluate the prevalence and predictors of Occult HCV among hemodialysis (HD) patients who achieved 24 weeks sustained virological response (SVR) after treatment with direct-acting antiviral agents (DAA) by detection of viral RNA in their peripheral blood mononuclear cells.

DETAILED DESCRIPTION:
In maintenance hemodialysis (MHD) patients, hepatitis C virus (HCV) infection is common and may be associated with poor clinical outcomes. A lot of treatment options for HCV have rapidly evolved over the past 5 years and various treatment choices for patients with advanced CKD are currently available.1 The reappearance of HCV infection months or years after sustained virologic response (SVR) may be due to the persistence of HCV in tissue cells in spite of being undetected in serum. This situation is known as occult hepatitis C infection (OCI).2 OCI is now a challenging entity in the field of post hepatitis management and follow-up. OCI is described when HCV-RNA is detectable in liver and/or peripheral blood mononuclear cells (PBMCs) in patients with undetectable serum HCV-RNA. To our knowledge , this is the first research to issue this problem in dialysis patients after treatment with direct acting antiviral drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients on regular hemodialysis treatment for more than 6 months.
* Achieved sustained virological response 24 weeks after the end of treatment with directly acting antiviral drugs (DAADs).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Occult HCV infection | 6 months
  By assessing presence of HCV RNA in peripheral blood mononuclear cells (PBMCs)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — Lecturer of Nephrology & Internal Medicine, Faculty of medicine, Alexandria University; Shady F Abouelnaga, MD, Study Chair — fellow of Clinical and Chemical Pathology Department, Alexandria University Hospitals; Hend N Abd Elmoteleub, MD, Study Chair — Lecturer of Hepatolgy and Internal Medicine Department, Faculty of Medicine, Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Maduell F, Belmar L, Ugalde J, Laguno M, Martinez-Rebollar M, Ojeda R, Arias M, Rodas L, Rossi F, Llovet LP, Gonzalez LN, Mallolas J, Londono MC. Elimination of hepatitis C virus infection from a hemodialysis unit and impact of treatment on the control of anemia. Gastroenterol Hepatol. 2019 Mar;42(3):164-170. doi: 10.1016/j.gastrohep.2018.07.015. Epub 2018 Oct 4. English, Spanish. PMID 30293914
- [Background] Naghdi R, Ranjbar M, Bokharaei-Salim F, Keyvani H, Savaj S, Ossareh S, Shirali A, Mohammad-Alizadeh AH. Occult Hepatitis C Infection Among Hemodialysis Patients: A Prevalence Study. Ann Hepatol. 2017 Jul-Aug;16(4):510-513. doi: 10.5604/01.3001.0010.0277. PMID 28611267
- [Derived] Naguib H, Abouelnaga SF, Elsayed MM. Occult hepatitis C virus infection in hemodialysis patients who achieved a sustained virological response to directly acting antiviral drugs: is it a concern? Int Urol Nephrol. 2024 Jan;56(1):217-222. doi: 10.1007/s11255-023-03621-1. Epub 2023 May 20. PMID 37209238